CLINICAL TRIAL: NCT01032668
Title: The EFFect of hIgh Dose ClopIdogrel treatmENT in Patients With Clopidogrel Resistance
Acronym: EFFICIENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BYİEAH2
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention, clopidogrel resistance, ASA resistance
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high dose clopidogrel (Experimental)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — high dose clopidogrel continuing after percutaneous coronary intervention

SUMMARY:
Continuing high dose clopidogrel treatment after elective PCI decreased adverse cardiac events in patients with clopidogrel resistance

DETAILED DESCRIPTION:
Aim:

Primary objective:

* To evaluate the effect of continuing high dose clopidogrel treatment on adverse cardiac events after elective PCI in patients with clopidogrel resistance

Secondary objective:

* To evaluate the effect of continuing high dose clopidogrel treatment on adverse cardiac events after elective PCI
* To evaluate the effect of continuing high dose clopidogrel treatment on bleeding complications after elective PCI
* To evaluate the clinical effect of VerifyNow which use as a clopidogrel resistance kit.

Study central:

Bursa Postgraduate Hospital, Cardiology Clinic

Study population:

we planned to enrol 180 patients. 50% of patients without clopidogrel resistance (control group: 90 patients) 50% have clopidogrel resistance. Than we randomise the patients (with clopidogrel resistance) in two groups (group 1:45 patients (75mg/day), group 2:45 patients (150mg/day))

inclusion criteria:

* The patients; who have planned elective PCI and have had written informed consent for participation to study.
* Age>18 year-old,
* The native coronary artery;lesion with narrowing >=70%

Exclusion criteria:

* Patients have allergy for ASA, Clopidogrel and heparin
* Patients who performed primary PCI
* Patients with acute coronary syndrome
* Patients with have a history of PCI and use clopidogrel
* Patients on warfarin therapy
* Patients who have bleeding diathesis, or have high risk for bleeding.

Study works:

* Write case report form for all patients
* Control for inclusion criteria.
* Evaluate the clopidogrel and ASA resistance with VerifyNow kit. Than randomised the patients.
* Demographic data (age, gender)
* Height, weight, BMI and GFR
* Risk factors
* laboratory data (biochemical and hematologic)
* Medication history
* Echocardiographic data
* Angiographic data
* PCI data(vessel diameter, stent diameter, lesion and stent length, performed PTCA or not, etc)
* Note complication (MACE, bleeding, hematoma etc)

  4 weeks later note the first control data and re assess the clopidogrel resistance with VerifyNow kit in patients groups 1 and 2.

Six months later note the second control data.

ELIGIBILITY:
Inclusion Criteria:

* The patients; who have planned elective PCI and have had written informed consent for participation to study.
* Age>18 year-old,
* The native coronary artery;lesion with narrowing >=70%

Exclusion Criteria:

* Patients have allergy for ASA, Clopidogrel and heparin
* Patients who performed primary PCI
* Patients with acute coronary syndrome
* Patients with have a history of PCI and use clopidogrel
* Patients on warfarin therapy
* Patients who have bleeding diathesis, or have high risk for bleeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Death, MI, TVR revascularization, stroke (MACCE) within 30 days and 6 moths | 6 months.

SECONDARY OUTCOMES:
Major or minor bleeding according to TIMI criteria 30 days and 6 months To evaluate the clinical effect of VerifyNow which use as a clopidogrel resistance kit 30 days and 6 months. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hasan ARI, MD, Study Director — Bursa Postgraduate Hospital
Locations (1):
- Bursa Yüksek İhtisas Eğitim ve Araştırma Hastanesi, Bursa, Turkey (Türkiye)

REFERENCES:
- [Background] Aleil B, Jacquemin L, De Poli F, Zaehringer M, Collet JP, Montalescot G, Cazenave JP, Dickele MC, Monassier JP, Gachet C. Clopidogrel 150 mg/day to overcome low responsiveness in patients undergoing elective percutaneous coronary intervention: results from the VASP-02 (Vasodilator-Stimulated Phosphoprotein-02) randomized study. JACC Cardiovasc Interv. 2008 Dec;1(6):631-8. doi: 10.1016/j.jcin.2008.09.004. PMID 19463377
- [Derived] Ari H, Ozkan H, Karacinar A, Ari S, Koca V, Bozat T. The EFFect of hIgh-dose ClopIdogrel treatmENT in patients with clopidogrel resistance (the EFFICIENT trial). Int J Cardiol. 2012 Jun 14;157(3):374-80. doi: 10.1016/j.ijcard.2010.12.083. Epub 2011 Jan 15. PMID 21239075